CLINICAL TRIAL: NCT04067661
Title: A Couples-Based Approach to HIV Prevention for Transgender Women and Their Male Partners
Brief Title: A Couples-based Intervention for Transgender Women and Their Partners
Acronym: T2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: NIH terminated funding for this project stating "This award no longer effectuates agency priorities."
Sponsor: University of Michigan (Other)
Collaborators: University of California, San Francisco (Other); Emory University (Other); Research Foundation for Mental Hygiene, Inc. (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kristi Gamarel, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: F050837; 5R01MH115765-05 (NIH)
Record Dates: First submitted 2019-08-22; First posted 2019-08-26 (Actual); Results first posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: HIV Infections; HIV Primary Infection
Keywords: HIV Prevention; Transgender Women; Intervention
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: The study involved a randomized controlled trial comparing the couples-based HIV prevention to an enhanced standard of care control condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants and their partners will complete four couples counseling sessions focused on developing and enhancing relationship skills to decrease HIV risk behaviors.
  Interventions: Behavioral: CHIP
- Control (Active Comparator): Participants and their partners will receive information and referrals on HIV risk and prevention strategies.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: CHIP — The couples-based HIV prevention intervention consists of four couples counseling sessions focused on relationship skills to decrease HIV risk behaviors.
  Other Names: It Takes Two
  Arms: Intervention
Behavioral: Control — Enhanced standard of care, which includes information and referrals on HIV risk and prevention.
  Arms: Control

SUMMARY:
This project seeks to test the efficacy of a couples-based HIV prevention program in large-scale randomized controlled trial (RCT) to reduce HIV risk among transgender woman and their partners. This project involves enrolling a racially diverse sample of transgender women and their partners and randomizing 50 couples to either the couples-based HIV prevention intervention or an enhanced standard of care (SOC) control condition. Couples will be followed quarterly over 12-months. Analysis of study outcomes will utilize both individual- and dyadic-level data. The primary outcome is a composite measure of risk for HIV transmission which encompasses validated behavioral indicators of HIV risk as well as biomedical confirmation of viral suppression and PrEP adherence.

DETAILED DESCRIPTION:
Transgender women (trans women; individuals with a feminine and/or female gender identity who were assigned male at birth) are disproportionately affected by HIV. One of the most consistently reported contexts for HIV transmission among trans women is within a primary partnership. In this partnership context, trans women report low condom use, difficulty disclosing their HIV status and negotiating HIV prevention strategies, poor communication about whether they permit sex outside of the relationship, and low rates of routine HIV testing. Likewise, research among males who have sex with trans women has found high HIV prevalence, inconsistent condom use with trans women, and low engagement with HIV prevention services.

For the past 10 years the investigators have conducted research to identify intervention targets for reducing HIV transmission in trans women and their partner using qualitative, survey, and intervention adaptation methodologies. Based on these conceptual and empirical understandings of HIV transmission in these dyads, the investigative team developed and pilot tested the first known couples-based HIV prevention program for trans women and primary partners (called "Couples HIV Intervention Program" or CHIP). CHIP was feasible, acceptable, and produced significant reductions in condomless sex acts with primary and casual partners and in number of casual partners at 3-month follow-up compared to a control group.

The project seeks to test the efficacy of the CHIP intervention on reductions in a Composite Risk for HIV (CR-HIV) outcome. CR-HIV is a binary indicator of couple HIV risk using validated measures of sexual behavior (defined as condomless anal or vaginal sex with a serodiscordant or unknown HIV status primary or outside partner), as well as PrEP use among HIV-negative participants and viral suppression among HIV-positive partners. The study involves two-arm prospective RCT in which 50 trans women and their partners (100 participants) will complete a Baseline assessment and then complete assessments every 3 months for 12 months. Recruitment and study activities will occur in San Francisco, California.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Self-report that they are in emotional and/or sexual relationship for at least three months
* One partner must identify as a trans women (assigned the male gender at birth but identify as female or as a trans woman)
* Both partners must have engaged in condomless sex within the past 6 months with any partner
* Able to provide informed consent
* Speak and read English

Exclusion Criteria:

* Currently psychotic, suicidal, or manic
* Either partner reports that participating in the study would cause them physical harm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Stein, Study Director — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
We will compile structured de-identified datasets and can make them available for additional/secondary data analyses. For data sharing, the research team will follow the "standards for privacy of individually identifiable health information." Participants' records and results will not be identified. No contact information will be included in any archived datasets.

REFERENCES:
- [Result] Gamarel KE, Chakravarty D, Neilands TB, Hoff CC, Lykens J, Darbes LA. Composite Risk for HIV: A New Approach Towards Integrating Biomedical and Behavioral Strategies in Couples-Based HIV Prevention Research. AIDS Behav. 2019 Jan;23(1):283-288. doi: 10.1007/s10461-018-2229-8. PMID 30003506
- [Result] Sevelius JM, Gutierrez-Mock L, Zamudio-Haas S, McCree B, Ngo A, Jackson A, Clynes C, Venegas L, Salinas A, Herrera C, Stein E, Operario D, Gamarel K. Research with Marginalized Communities: Challenges to Continuity During the COVID-19 Pandemic. AIDS Behav. 2020 Jul;24(7):2009-2012. doi: 10.1007/s10461-020-02920-3. No abstract available. PMID 32415617
- [Result] Gamarel KE, Sevelius JM, Neilands TB, Kaplan RL, Johnson MO, Nemoto T, Darbes LA, Operario D. Couples-based approach to HIV prevention for transgender women and their partners: study protocol for a randomised controlled trial testing the efficacy of the 'It Takes Two' intervention. BMJ Open. 2020 Oct 15;10(10):e038723. doi: 10.1136/bmjopen-2020-038723. PMID 33060086

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 104 individuals (52 couples) were enrolled in the study.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 52 (26 transgender women participants and 26 partners in the "Intervention Arm" for a total of 52 individuals (26 dyads) randomized to the "Intervention Arm") | 52 (26 transgender women participants and 26 partners in the "Control Arm" for a total of 52 individuals (26 dyads) randomized to the "Control Arm")
Completed | 42 (21 transgender women participants and 21 partners in the "Intervention Arm" for a total of 42 individuals (21 dyads) completed the "Intervention Arm") | 50 (25 transgender women participants and 25 partners in the "Control Arm" for a total of 50 individuals (25 dyads) completed the "Control Arm")
Not Completed | 10 | 2

BASELINE CHARACTERISTICS:
Population: 104 individuals (52 couples) were enrolled; the results are presented at the individual-level. Since participants were recruited as dyads, tests for differences in baseline characteristics between intervention and control conditions were adjusted for non-independence in the data due to clustering at the couple level.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (1.8) | 35.5 (2.1) | 36.0 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 36 | 74
  Male | 14 | 16 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 6 | 20
  Not Hispanic or Latino | 37 | 45 | 82
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 7 | 7 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 9 | 14
  White | 29 | 24 | 53
  More than one race | 5 | 7 | 12
  Unknown or Not Reported | 5 | 4 | 9
Region of Enrollment [Number; unit: participants] — California
  participants
    United States | 52 | 52 | 104
Condomless sex [Count of Participants; unit: Participants] | 52 | 52 | 104

OUTCOME MEASURES:

1. Primary Outcome: Condomless Sex
Description: Self-report condomless anal or vaginal sex with any partner in the past 3 months
Time Frame: Changes in self-reported condomless anal or vaginal sex at 12-month follow-up
Population: We analyzed data at the individual level. The number presented represents that participants who competed their 12-month follow-up. Since participants were recruited as dyads, tests for differences in outcomes between intervention and control conditions were adjusted for non-independence in the data due to clustering at the couple level.
Measure: Number; unit: participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 42 | 50
participants | 20 | 31

2. Primary Outcome: Composite HIV Risk
Description: We created a composite measure incorporating self-reported condomless sex, PrEP adherence, and viral suppression, resulting in a binary HIV risk outcome (1=yes, 0=no). Participants reporting condomless sex in the past 30 days, along with either lack of viral suppression or non-adherence to PrEP, were categorized as at HIV risk. Conversely, those who did not report condomless sex, were virally suppressed, or were adherent to PrEP were placed in the not at HIV risk group. The variable was constructed such that 1= HIV Risk versus 0 = No HIV Risk. The results below represent the number of participants who were categorized as 1 = HIV risk at the 12-month follow up.
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 42 | 50
Participants | 17 | 28

ADVERSE EVENTS:
Time Frame: One year
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 0/52 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-12): https://cdn.clinicaltrials.gov/large-docs/61/NCT04067661/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-12): https://cdn.clinicaltrials.gov/large-docs/61/NCT04067661/ICF_001.pdf